CLINICAL TRIAL: NCT02580500
Title: Epidural and Spinal Anesthesia Techniques in Pilonidal Dermoid Sinus Surgeries: Prospective Randomized Trials
Brief Title: Epidural and Spinal Anesthesia Techniques in Pilonidal Dermoid Sinus Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lütfiye Nuri Burat Government Hospital (Other Government)
Responsible Party: Principal Investigator, TURGUT DONMEZ, General Surgeon, MD, Lütfiye Nuri Burat Government Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: lutfiye01
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Sinus; Dermal, Pilonidal
Keywords: Epidural anesthesia; Spinal anesthesia; pilonidal dermoid sinus
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): Pilonidal dermoid cyst surgery in Spinal anaesthesia
  Interventions: Procedure: spinal catheter
- group 2 (Active Comparator): Pilonidal dermoid cyst surgery in Epidural anaesthesia
  Interventions: Procedure: epidural catheter

INTERVENTIONS:
Procedure: epidural catheter — epidural anaesthesia application for spinal catheter will be used
  Arms: group 2
Procedure: spinal catheter — spinal anesthesia application for spinal catheter will be used
  Arms: group 1

SUMMARY:
Pilonidal dermoid cyst surgery under general anesthesia and regional anesthesia techniques is used.regional anesthesia techniques; spinal, epidural, spinal epidural (combined) and is the local anesthesia.In the investigators study, pilonidal dermoid cyst surgery in spinal and epidural anesthesia techniques activity, reliability will be compared to the side effects and complications.

One hundred patients will be randomly assigned to either the pilonidal dermoid cyst under Spinal anaesthesia (50 patients)(Group 1) or pilonidal dermoid cyst under epidural anaesthesia (50 patients)(Group 2). Group 1 will be used in spinal catheter in spinal anesthesia procedures or Group 2 will be used epidural catheter in epidural anaesthesia procedures.All patients has symptomatic pilonidal dermoid cyst.

DETAILED DESCRIPTION:
Pilonidal dermoid is a tubular skin defect which can be seen in both female and male patients between the ages of 12 to 80. Treatment alternatives includes surgical excision. During the surgical treatment local, general, spinal or epidural anesthesia could be applied. However, local anesthesia usually is not preferred due to the fact that pilonidal dermoid sinuses depth, width could not be determined precisely. General anesthesia also is not preferred due to the fact that difficulties arising from patient's positioning and positioning based potential lung related problems. In general, spinal anesthesia and epidural anesthesia is preferred for pilonidal dermoid sinus surgeries. In this study, the investigators will demonstrate advantages, disadvantages, complications, (sensory and motor block levels), and durations of spinal and epidural anesthesia and superiority of each on these subjects.

Patients who are over 18 and have a America Society of Anesthesiologist (ASA) physical score of I and II will be included in the study. Patients who are pregnant, have a known allergic reactions to local anesthetic and have contraindications against spinal and epidural anesthetic will be excluded from the study.

In this study the investigators separate the patients into 2 groups. Group1: pilonidal dermoid cyst under Spinal anaesthesia (50 patients).Group 1 will be used in spinal catheter in spinal anesthesia procedures ; Group2:pilonidal dermoid cyst under epidural anaesthesia (50 patient).Group 2 will be used epidural catheter in epidural anaesthesia procedures. All patients has symptomatic pilonidal dermoid cyst

ELIGIBILITY:
Inclusion Criteria:

* America Society of Anesthesiologist (ASA) physical score of I and II
* the men and women over the age of 18, pilonidal sinus disease

Exclusion Criteria:

* Pediatric patients
* Pregnant women
* Patients with bleeding disorder
* Patients with spinal deformity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
sensory block duration(time:hour) | up to 6 hours
  group1 and group 2

SECONDARY OUTCOMES:
Duration of operation(time:hour) | up to 2 hours
  group1 and group 2
Headache | from end of the operation to postoperative 3 days
  group 1 and group 2(participants)
Nausea/Vomiting | from end of the operation to postoperative 1 day
  group 1 and group 2(participants)
Urinary Retention | from end of the operation to postoperative 1 day
  group 1 and group 2 (participants)

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Donmez, Surgeon, Principal Investigator — Lutfiye Nuri Burat Goverment Hospital
Locations (1):
- Lutfiye NBGH, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Muslu B, Usta B, Muslu S, Yesilay A, Gozdemir M, Sert H, Demircioglu R. Effect of locally administered lornoxicam in the management of low back pain after lumbar epidural anesthesia: a double-blind, randomized, controlled study. Minerva Anestesiol. 2009 Sep;75(9):494-7. Epub 2009 May 21. PMID 19461565
- [Background] Orhon ZN, Koltka EN, Devrim S, Tufekci S, Dogru S, Celik M. Epidural anesthesia for pilonidal sinus surgery: ropivacaine versus levobupivacaine. Korean J Anesthesiol. 2015 Apr;68(2):141-7. doi: 10.4097/kjae.2015.68.2.141. Epub 2015 Mar 30. PMID 25844132